CLINICAL TRIAL: NCT04022031
Title: Prospective Cohort Study on Adjuvant Treatment of Coronary Heart Disease Angina Pectoris With Chinese Patent Medicine
Brief Title: Clinical Study on Adjuvant Treatment of Coronary Heart Disease Angina Pectoris With Chinese Patent Medicine
Acronym: CSCD-TCM
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Tianjin University of Traditional Chinese Medicine (Other)
Responsible Party: Principal Investigator, Chunquan Yu, researcher, Tianjin University of Traditional Chinese Medicine
Other Study IDs: CSCD-TCM
Record Dates: First submitted 2019-07-13; First posted 2019-07-16 (Actual); Last update posted 2019-07-17 (Actual); Status verified 2019-07

CONDITIONS: Atherosclerotic Heart Disease With Angina Nos

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood, urine, feces, tongue coating
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Exposed group: Chinese patent medicine combined with western medicine routine
  Interventions: Drug: Chinese patent medicine
- Non-exposed group: Western medicine routine treatment

INTERVENTIONS:
Drug: Chinese patent medicine — Shexiang Baoxin Pill, Tongxinluo Capsule, Tongmai Yangxin Pill, Xuefu Zhuyu Capsule, Qishen Yiqi Dropping Pill.
  Groups: Exposed group

SUMMARY:
A prospective cohort study was performed in patients with angina pectoris who were treated with oral Chinese patent medicine and Western medicine.Collect primary and secondary efficacy indicators such as the incidence of cardiovascular events, using clinical samples to detect genomics, proteomics, metabolomics, intestinal flora and sclerotia.To explore the clinical efficacy of Chinese patent medicine in the treatment of coronary heart disease with angina pectoris, and provide reliable data support for its clinical application.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily participate, understand and sign the informed consent form;
2. Age 35-75 years old, gender is not limited;
3. Patients with coronary heart disease and angina pectoris in the Department of Cardiology or Outpatient Department, the diagnosis of angina pectoris meets the diagnostic criteria of Western medicine and the standard of TCM syndrome differentiation;
4. Patients who met the criteria for drug treatment, the exposed group was treated with traditional Chinese medicine combined with Western medicine, and the non-exposed group was treated with Western medicine alone.

Exclusion Criteria:

1. Combined with other heart diseases, neurosis, menopausal syndrome, hyperthyroidism, cervical or vertebral artery type cervical spondylosis, gastro-oesophageal reflux disease or esophageal hiatus hernia may cause chest pain;
2. Patients with severe symptoms and uncontrollable angina pectoris, with acute myocardial infarction, heart failure, myocarditis, cardiomyopathy, severe heart valve disease, liver failure or renal failure, malignant tumors and serious metabolic diseases;
3. Pregnant women, lactating women or women of childbearing age who have birth requirements;
4. Mental patients, or cognitive dysfunction;
5. Participated in other clinical trials in the last 3 months;
6. Allergic persons, or those known to be allergic to therapeutic drugs;
7. It is expected that the compliance is poor and it is not possible to visit regularly;
8. Patients who do not have a current address or whose current address is incomplete and have no contact number;
9. The investigator believes that there are other situations that are not suitable for the trial.

Ages: 35 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The collaboration network of coronary heart disease research medical units formed by the research group, including the First Affiliated Hospital of Tianjin University of Traditional Chinese Medicine, the Second Affiliated Hospital of Tianjin University of Traditional Chinese Medicine, Tianjin Chest Hospital, Tianjin Nankai Hospital, Tianjin Medical University General Hospital，a total of 5 hospitals.
Sampling Method: Non-Probability Sample
Enrollment: 12400 (Estimated)
Dates: Start 2019-09-01 (Estimated); Primary Completion 2021-09-01 (Estimated); Study Completion 2022-09-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of cardiovascular events | one year
  These include acute myocardial infarction (AMI), percutaneous coronary intervention (PCI), or coronary artery bypass grafting (CABG).

SECONDARY OUTCOMES:
Death from all causes | one year
Re-admission due to cardiovascular events | one year
Seattle Angina Questionnaire | three months
Clinical biochemical test | three months
Film degree exam | three months

CONTACTS AND LOCATIONS:
Locations (1):
- Tianjin University of Traditional Chinese Medicine, Tianjin, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: Yes